CLINICAL TRIAL: NCT03123328
Title: Evaluation of Non-Invasive Hemoglobin in Trauma Patients Using FDA-Cleared Masimo Pulse CO-Oximeter
Brief Title: Evaluation of Non-Invasive Hemoglobin in Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HOLC0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subjects (Experimental): Each test subject will receive a Radical-7 Pulse CO-Oximeter and sensor that will remain on the subject for the first 24 hours following ED admission or discharge from the ICU/IMU.
  Interventions: Device: Radical-7 Pulse CO-Oximeter and sensor

INTERVENTIONS:
Device: Radical-7 Pulse CO-Oximeter and sensor — Noninvasive device that measures hemoglobin.

SUMMARY:
This is a prospective, non-blinded, non-randomized, interventional study of the Masimo pulse oximeter and sensors in a trauma setting

DETAILED DESCRIPTION:
The study aimed to evaluate SpHb's ability to detect critical drops in a trauma population

ELIGIBILITY:
Inclusion Criteria:

* Estimated 16 years of age or older or greater than or equal to 50 kg body weight if age unknown.
* Level 1 (highest trauma activation) status at the time of arrival to emergency department (ED).
* Expected to be admitted to the ICU/IMU for in hospital care.

Exclusion Criteria:

* Moribund patients with devastating injuries and expected to die within one hour of ED admission.
* Prisoners, as defined as those who have been directly admitted from a correctional facility (a free living individual who is under police observation as a suspect will remain in the study until hospital discharge).
* Obvious pregnancy in the ED.
* Received greater than 5 minutes of cardiopulmonary resuscitation (CPR) in the pre-arrival or hospital setting.
* Has, on the ring, middle and index fingers of both hands, any of the following: finger deformities, injuries, including burns, scar tissue or infection, or any material that may interfere with sensor application or trans-illumination of the site.
* Has significant bilateral trauma to the arms or forearms.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Subjects
Started | 380
Completed | 351
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects
Number analyzed (Participants) | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 294
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 281
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 7
  Race/Ethnicity: Black or African American | 95
  Race/Ethnicity: White | 152
  Race/Ethnicity: More than one race | 1
  Race/Ethnicity: Unknown or Not Reported | 3
  Race/Ethnicity: Hispanic/Latino | 92
  Race/Ethnicity: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: SpHb's Ability to Detect Critical Drops
Description: The ability of noninvasive continuous total hemoglobin (SpHb) to detect critical drops in arterial or venous hemoglobin values, calculated using chi-squared analysis.
Time Frame: Up to 24 hours.
Population: Sufficient number of cases to meet sample size criteria for assessing outcomes was not achieved. The protocol required a minimum of 50 subjects with at least 2 blood samples to conduct an interim analysis to calculate final sample size in order to obtain to a definition of critical drop detection. This study was not able to meet this target and therefore a critical drop could not be defined (primary outcome measure).
Arm/Group | Test Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored during participation in the study in the ED and their stay in ICU.
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 1/351
Serious Adverse Events (participants affected / at risk) | 0/351
Other Adverse Events (participants affected / at risk) | 0/351

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03123328/Prot_SAP_000.pdf